CLINICAL TRIAL: NCT04408222
Title: Awake Proning in Patients With COVID-19-Induced Acute Hypoxemic Respiratory Failure
Brief Title: Awake Proning in COVID-19 Patients With Hypoxemic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sanja Jelic, Associate Professor of Medicine, Columbia University
Other Study IDs: AAAT0134
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Oxygen Deficiency; Coronavirus Infection
Keywords: Awake Proning; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Hypoxia; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Awake Proning: COVID-19 patients with hypoxemic respiratory failure with awake prone positioning, as tolerated, up to 24 hours daily.
  Interventions: Other: Awake proning

INTERVENTIONS:
Other: Awake proning — Prone positioning of awake, as tolerated, for up to 24 hours daily.

SUMMARY:
The purpose of this study is to retrospectively review clinical data to determine whether awake proning improves oxygenation in spontaneously breathing patients with COVID-19 severe hypoxemic respiratory failure.

DETAILED DESCRIPTION:
Critically ill patients with coronavirus disease 2019 (COVID-19) severely strained intensive care resources in New York in April 2020. The prone position improves oxygenation in intubated patients with acute respiratory distress syndrome. The investigators wanted to study whether the prone position is associated with improved oxygenation and decreased risk for intubation in spontaneously breathing patients with severe COVID-19 hypoxemic respiratory failure. Awake prone positioning was implemented based on the health care provider decision.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to the Columbia University step-down unit from April 6, 2020.
* Laboratory confirmed COVID-19 infection with severe hypoxemic respiratory failure defined as respiratory rate ≥30 breaths/min and oxyhemoglobin saturation (SpO2) ≤93% while receiving supplemental oxygen 6 L/min via nasal cannula and 15 L/min via non-rebreather facemask.

Exclusion Criteria:

* Altered mental status with inability to turn in bed without assistance
* Extreme respiratory distress requiring immediate intubation, or oxygen requirements less than specified in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with laboratory-confirmed COVID-19 infection who were admitted to the step-down unit at the Columbia University Irving Medical Center in New York between April 6 and 14, 2020 were included. A confirmed case of COVID-19 was defined by a positive result on a reverse transcriptase-polymerase chain reaction (RT-PCR) assay of a specimen collected on a nasopharyngeal swab. Only laboratory-confirmed cases were included.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Change in SpO2 | Before proning and 1 hour after initiation of the prone position
  SpO2 was measured by peripheral pulse oximetry.

SECONDARY OUTCOMES:
Mean Risk Difference in Intubation Rates | Duration of hospitalization or up to 1 month from admission
  The mean risk difference in intubation rates for patients with SpO2 ≥95% vs. <95% 1 hour after initiation of the prone position was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Jelic, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared owing to privacy protection.

REFERENCES:
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414
- [Background] Sun Q, Qiu H, Huang M, Yang Y. Lower mortality of COVID-19 by early recognition and intervention: experience from Jiangsu Province. Ann Intensive Care. 2020 Mar 18;10(1):33. doi: 10.1186/s13613-020-00650-2. No abstract available. PMID 32189136
- [Background] Perez-Nieto OR, Guerrero-Gutierrez MA, Deloya-Tomas E, Namendys-Silva SA. Prone positioning combined with high-flow nasal cannula in severe noninfectious ARDS. Crit Care. 2020 Mar 23;24(1):114. doi: 10.1186/s13054-020-2821-y. No abstract available. PMID 32204726
- [Background] Ding L, Wang L, Ma W, He H. Efficacy and safety of early prone positioning combined with HFNC or NIV in moderate to severe ARDS: a multi-center prospective cohort study. Crit Care. 2020 Jan 30;24(1):28. doi: 10.1186/s13054-020-2738-5. PMID 32000806
- [Background] https://www1.nyc.gov/site/doh/Covid/Covid-19-data.page; Accessed April 17, 2020.